CLINICAL TRIAL: NCT05605197
Title: Clinical Study to Evaluate the Safety and Efficacy of U87 CART in Treatment of Advanced Solid Tumor
Brief Title: U87 CART in Treatment of Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U87-3
Record Dates: First submitted 2022-10-03; First posted 2022-11-04 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer; Solid Tumor, Adult
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- U87 CAR-T cells (Experimental): The Patients are enrolled into 2 dose level cohorts in sequence
  Interventions: Drug: U87 CAR-T

INTERVENTIONS:
Drug: U87 CAR-T — Subjects will be pretreated with cyclophosphamide 250~500 mg/m2( body surface area) for 3 days prior to Intravenous injection of U87, followed by intraartery of U87 14 days later with intravenous IL-2. Researchers can perform intratumoral injection based on their judgment.This study will explore two dose of dose 1 (DL-1): 1×106 (±20%) to dose 2 (DL-2): 1×107 (±20%),each group was enrolled in 3~6 patients.

SUMMARY:
This is a single center, open-label, phase 1 study to evaluate the safety and efficacy of U87 CART in treating advanced solid tumor .

DETAILED DESCRIPTION:
Following consent, patients must have tumor tissue evaluated by IHC assay. Patients meeting all eligibility criteria will undergo a leukapheresis procedure to collect autologous mononuclear cells for manufacture of investigational drug product (U87). Following manufacture of the drug product, subjects will receive preconditioning prior to U87 infusion. All subjects will be asked to continue to undergo long-term gene safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary informed consent is given;
2. Age 18 to 75;
3. Patients with pathologically confirmed advanced solid tumor who have failed first-line therapy; or patients who are intolerant to first-line standard therapy and voluntarily give up standard therapy;
4. Immunohistochemical (IHC) staining of tumor tissue samples from patients was positive for U87 specific antigen (≥ 2 +, and the expression rate was ≥ 20%);
5. Expected survival ≥12 weeks;
6. Measurable tumor lesions according to RECIST 1.1;
7. ECOG performance score 0-1;
8. Sufficient venous access for mononuclear cell collection;
9. HBc Ab positive, HBsAg negative can be included in the group when the PCR detection of HBV DNA is negative;
10. Patients should maintain adequate organ function;
11. Dyspnea (CTCAE v5.0) ≤ Grade 1; Blood oxygen saturation>91% without oxygen inhalation;
12. Pregnancy test was negative in women of childbearing age; Both male and female subjects should agree to use effective contraceptives during the treatment period and within the following year;

Exclusion Criteria:

1. Pregnant or lactating women;
2. Uncontrolled active infections;
3. Active Syphilis, HIV, hepatitis B or hepatitis C infection;
4. Congenital immunodeficiency;
5. Have serious allergic reaction to any drug to be used in this study;
6. Other incurable malignant tumors in the past three years;
7. History or presence of clinically relevant CNS pathology such as epilepsy, Cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any CNS-related autoimmune disease;
8. Have undergone cardiac angioplasty or stent implantation within 12 months, or have a history of myocardial infarction, unstable angina or other clinically significant heart diseases;
9. Subjects requiring anticoagulation or long-term antiplatelet therapy;
10. Subjects who have undergone major surgery or significant trauma within four weeks before enrolled in the study.
11. Other situations that the investigator thinks are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after U87 CAR-T cells infusion [Safety and Tolerability] | 28 days post administration of CAR-T-cells
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0) Dose-limiting toxicity after U87 CAR-T cells infusion.

SECONDARY OUTCOMES:
Disease control rate (DCR) of U87 CAR-T cells treatment in advanced solid tumor. [Effectiveness] | 2 years post CAR T cell infusion
  Disease control rate: including CR, PR and SD(Assessed based on RECIST 1.1 criteria)
Objective response rate (ORR) of U87 CAR-T cells treatment in advanced solid tumor. [Effectiveness] | 2 years post CAR T cell infusion
  Objective response rate includes：CR、PR(Assessed based on RECIST1.1 criteria)
Duration of Response (DOR) of U87 CAR-T cells treatment in advanced solid tumot[Effectiveness] | 2 years post CAR T cell infusion
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of U87 CAR-T cells treatment in advanced solid tumor[Effectiveness] | 2 years post CAR T cell infusion
  PFS will be assessed from the first U87 CAR-T cells infusion to death from any cause or the first assessment of progression(Assessed based on RECIST1.1 ） criteria)
Overall survival(OS) of U87 CAR-T cells treatment in advanced solid tumor [Effectiveness] | 2 years post CAR T cell infusion
  OS will be assessed from the first U87 CAR-T cells infusion to death from any cause (Assessed based on RECIST 1.1 criteria)
Pharmacokinetics of U87 CAR-T cells | 2 years post CAR T cell infusion
  Peak value of eripheral blood (Cmax)
Pharmacokinetics of U87 CAR-T cells | 2 years post CAR T cell infusion
  Area under the eripheral blood concentration versus time curve (AUC)
Pharmacokinetics of U87 CAR-T cells | 2 years post CAR T cell infusion
  Time of peak value
Pharmacodynamics of U87 CAR-T cells | 2 years post CAR T cell infusion
  Concentration levels of CAR-T-related serum cytokines such as IL-6, IFN γ, IL-2, TNFα, ferritin and CRP at each time point

CONTACTS AND LOCATIONS:
Locations (1):
- China Shanghai 10th People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No